CLINICAL TRIAL: NCT03947749
Title: Linking Epigenomics With Prescription Opioid Abuse and High Impact Musculoskeletal Pain
Acronym: LEAP
Status: Completed | Type: Observational
Sponsor: University of Florida (Other)
Collaborators: Florida Medical Malpractice Joint Underwriting Association (Unknown)
Responsible Party: Sponsor
Other Study IDs: IRB201901297
Record Dates: First submitted 2019-05-09; First posted 2019-05-13 (Actual); Last update posted 2023-08-14 (Actual); Status verified 2023-08

CONDITIONS: Pain, Chronic; Prescription Drug Abuse (Not Dependent)
MeSH Terms: conditions — Chronic Pain; Substance-Related Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Mouthwash samples will be collected in all enrolled subjects
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Patients with HICMP: Patients with PROMIS Pain Interference-6b scores one standard deviation above the national average will be categorized into this group.
- Patients without HICMP: Patients without PROMIS Pain Interference-6b scores one standard deviation above the national average will be categorized will be categorized into this group.
- Patients at risk for opioid abuse or misuse: The Opioid Risk Tool and PROMIS Short Form v1.0-Prescription Pain Medication Misuse will be used to categorize patients at risk.
- Patients not at risk for opioid abuse or misuse: The Opioid Risk Tool and PROMIS Short Form v1.0-Prescription Pain Medication Misuse will be used to categorize patients at risk.

SUMMARY:
Genetic variability from epigenetic modification of genes related to pain physiology and opioid pharmacodynamics may influence susceptibility to high-impact chronic musculoskeletal pain, opioid efficacy, and vulnerability to opioid abuse. Exploring the role of epigenomics and opioid addiction may improve understanding and treatment of these complex multifactorial conditions and, potentially, reduce their development.

DETAILED DESCRIPTION:
Over 19 million adults suffer with chronic pain, which frequently limits life or work activities. Many of these patients are chronic prescription opioid consumers and may be at risk for opioid use disorder. Genetic variability of genes related to pain physiology and opioid pharmacodynamics may influence susceptibility to high-impact chronic musculoskeletal pain (HICMP), opioid efficacy, and vulnerability to opioid abuse. There is a paucity of research on the epigenetic profile of patients with HICMP and of those who fall in the spectrum between opioid addicted and opioid naive. Exploring the role of epigenomics in HICMP and opioid addiction may improve understanding and treatment of these complex multifactorial conditions and, potentially, reduce development.

The long-term goal is to create a profile of genetic and psychosocial risk factors for identifying patients susceptible to HICMP and opioid abuse. The objective of this pilot study is to gather preliminary data on the association of epigenetic modification of genes with HICMP and prescription opioid abuse.The study team propose to compare COMT and OPRM1 DNA methylation patterns in patients with HICMP (Group 1) to those without HICMP (Group 2).The investigators will also correlate OPRM1 DNA methylation patterns with the likelihood of misuse and abuse in chronic opioid consumers. It is hypothesized: (1) the promoter region of the COMT and OPRM1 genes will be hypo- and hyper-methylated, respectively, in Group 1 compared to Group 2; and (2) the OPRM1 gene in patients at high risk for opioid misuse and abuse will be hyper-methylated.

ELIGIBILITY:
Inclusion Criteria:

* Patients age ≥18 years with chronic musculoskeletal pain (pain present for 3 or more months) treated with prescription opioids on most days in the past 3 months.

Exclusion Criteria:

* Patients who are non-English speaking,
* Patients who are incarcerated
* Patients who are unable to provide consent will be excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study population will be adult patients with chronic musculoskeletal pain (pain present for 3 or more months) treated with prescription opioids on most days in the past 3 months.
Sampling Method: Non-Probability Sample
Enrollment: 275 (Actual)
Dates: Start 2019-09-25 (Actual); Primary Completion 2023-04-05 (Actual); Study Completion 2023-04-06 (Actual)

PRIMARY OUTCOMES:
PROMIS Pain Interference 6b | Baseline
  Symptom assessment tool measures six items on 5-point scales for pain interference on aspects of daily life. The higher the total score, the more severe the symptom.
Opioid Risk Tool | Baseline
  Prescription opioid abuse or misuse will be measured using the Opioid Risk Tool. This tool should be administered to patients upon an initial visit prior to beginning opioid therapy for pain management. A score of 3 or lower indicates low risk for future opioid abuse, a score of 4 to 7 indicates moderate risk for opioid abuse, and a score of 8 or higher indicates a high risk for opioid abuse.
PROMIS Short Form v1.0-Prescription Pain Medication Misuse | Baseline
  Seven question survey concerning prescription pain medication use within the last 3 months. Self reported answers ranging 1-5; with 1 being 'never' to 5 being 'almost always.' Prescription opioid abuse or misuse will be measured using the PROMIS Short Form v1.0-Prescription Pain Medication Misuse. Patients with PPMM scores of 60 or more will be considered high risk for opioid misuse or abuse.

CONTACTS AND LOCATIONS:
Overall Officials: Sophia Sheikh, MD, Principal Investigator — University of Florida
Locations (2):
- United States (2):
  - UF Health of University of Florida, Gainesville, Florida
  - UF Health - Jacksonville, Jacksonville, Florida

IPD SHARING:
Plan to Share IPD: No